CLINICAL TRIAL: NCT02304692
Title: C49:Clinical Survey of Different Abutment Topologies Installed With a Minimally Invasive Surgery for Bone Anchored Hearing Systems
Brief Title: Clinical Survey of Different Abutment Topologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C49
Record Dates: First submitted 2014-11-14; First posted 2014-12-02 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Conductive Hearing Loss; Unilateral Partial Deafness; Mixed Hearing Loss
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oticon Medical Machined Abutment (Sham Comparator): A non surface modified abutment is used
  Interventions: Device: Bone anchored hearing aid
- Oticon Medical Modified Abutment (Experimental): A surface modified abutment is used
  Interventions: Device: Bone anchored hearing aid

INTERVENTIONS:
Device: Bone anchored hearing aid
  Other Names: BAHS; BAHA

SUMMARY:
This study is designed to compare two different surfaces of bone anchored hearing aid abutments in terms of bacterial colonization, inflammatory response and skin reactions.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (18 years of age or older) patient eligible for a bone anchored hearing system

Exclusion Criteria:

* Inability or unwillingness to participate in follow-up
* Skin thickness of > 10 mm
* Diseases known to compromise bone quality
* Irradiated in the implant area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of colony forming units (CFU) | 3 months post-surgery
  The primary end point is CFU counts 3 months post-surgery.

SECONDARY OUTCOMES:
Number of colony forming units (CFU) on abutment (CFU/abutment) | 3 months post-surgery
Number of colony forming units (CFU) on abutment (CFU/abutment) | 12 months post-surgery
Number of colony forming units (CFU), strip (CFU/strip) | 3 months post-surgery
Number of colony forming units (CFU), strip (CFU/strip) | 12 months post-surgery
Number of colony forming units (CFU) in tissue samples (CFU/mg | 3 months post-surgery
Number of colony forming units (CFU) in tissue samples (CFU/mg | 12 months post-surgery
RNA level for host inflammatory response | 3 months post-surgery
RNA level for tissue repair | 3 months post-surgery
RNA level for host host microbial infection response | 3 months post-surgery
RNA level for host inflammatory response | 12 months post-surgery
RNA level for tissue repair | 12 months post-surgery
RNA level for host host microbial infection response | 12 months post-surgery
Histology investigation of tissue biopsy | 3 months post-surgery
Histology investigation of tissue biopsy | 12 months post-surgery

OTHER OUTCOMES:
Skin status according to Holgers and clinical assessment | 3 months post surgery
Skin status according to Holgers and clinical assessment | Up to 24 months post surgery
Postoperative complications | 3 months post surgery
Pain and numbness | Up to 24 months post surgery
Implant stability by clinical assessment and implant stability quotient (ISQ)measurements | Up to 24 months post surgery
Pocket depth | 6 months post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Jonhede, Study Chair — Sponsor GmbH
Locations (1):
- Department of Otorhinolaryngology, Karolinska University Hospital, Stockholm, Sweden